CLINICAL TRIAL: NCT03579329
Title: Effect of Total Knee Arthroplasty on Sarcopenia in Patients With Osteoarthritis in the Knee
Acronym: Sarcopenia
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Ho Ki Wai, Clinical Professional Consultant, Chinese University of Hong Kong
Other Study IDs: 2015.539
Record Dates: First submitted 2018-06-26; First posted 2018-07-06 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Sarcopenia; Osteoarthritis, Knee
Keywords: sarcopenia; Osteoarthritis; Total Knee Arthroplasty
MeSH Terms: conditions — Sarcopenia; Osteoarthritis, Knee; Osteoarthritis | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Total Knee Arthroplasty — Effect of Total Knee Arthroplasty on Sarcopenia in Patients with Osteoarthritis in the Knee

SUMMARY:
Sarcopenia is a wasting disease with the locomotion system in the aged population. It is defined as the decline in muscle mass (lean body mass) and strength with the advance of age. The prevalence of sarcopenia increases with age, reaching an astounding 50% among the population aged over 75 in the United States. Sarcopenia is often associated with frailty, falls, and disability. Studies have found sarcopenia can be a predicting risk factor for fractures in the elderly. In addition, sarcopenia predicted a higher chance of mortality in nursing homes.

DETAILED DESCRIPTION:
Notably, sarcopenia often accompanies with osteoarthritis (OA). However, the relationship between sarcopenia and OA is still unclear. One understanding is that sarcopenia and OA and co-existing conditions. One study identified sarcopenia as one of the risk factors of OA. There is also a study which speculated that OA may inhibit the progression of sarcopenia since they observed OA patients had higher BMP4-positive tissues, which indicated presence of satellites cells that may increase muscle regeneration capabilities.

However, more studies suggested that OA may contribute to the development of sarcopenia among the elderly. First, it is observed that the prevalence of sarcopenia among OA patients is higher than among the normal population. Further, cross-sectional studies demonstrated that hip or knee OA are associated with declines in muscle mass and muscle strength. Most interestingly, female patients with knee OA had declined lean body mass in their lower limbs, but not in their upper limbs or trunks.

Major risk factors of sarcopenia include malnutrition and lack of physical exercise. Therefore, diet supplementation and exercise potentially provide means to alleviate sarcopenia. Studies have demonstrated that strength training in the elderly can improve sarcopenia by increasing muscle strength, mass, power and quality. Exercise habit in middle age could prevent sarcopenia in elder age, maintaining better scores in grip strength, gait speed, and one-leg standing time. Possible molecular mechanism of exercise on sarcopenia is the upregulated nuclear factor-erythroid 2 p45-related factor 2 (Nrf2)-mediated antioxidant response cascade in skeletal muscle, which protected the muscle from oxygen species-mediated toxicity.

OA patients often adopt a sedentary life style to avoid joint pain and stiffness, which probably triggers the dysfunction of Nrf2 -mediated antioxidant response cascade, eventually leading to skeletal muscle atrophy. With the ultimate solution, total knee anthroplasty (TKA), patients with knee OA gradually regain their mobility and greatly increase their social and physical activities. Therefore, one can expect to see improved sarcopenia in patients with knee OA after TKA.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female aged over 18 wirh end stage knee OA
* Scheduled for TKA
* Agree to provide written consent

Exclusion Criteria:

* History of alcoholism or drug abuse
* Pregnancy and breast-feeding
* Presence of serious pathologies
* Steroid-based systemic therapy in progress or interrupted since less than 1 month
* With significant hematologic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: End stage knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | one year
  Questionnaire
DXA scan | one year
  Lean Muscle Mass Index

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | one year
  Questionnaire
Self-Rated 12 | one year
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopaedics & Traumatology, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ho KK, Lau LC, Chau WW, Poon Q, Chung KY, Wong RM. End-stage knee osteoarthritis with and without sarcopenia and the effect of knee arthroplasty - a prospective cohort study. BMC Geriatr. 2021 Jan 4;21(1):2. doi: 10.1186/s12877-020-01929-6. PMID 33397330